CLINICAL TRIAL: NCT04343885
Title: UpFrontPSMA : A Randomised Phase 2 Study of Sequential 177Lu-PSMA617 and Docetaxel Versus Docetaxel in Metastatic Hormone-Naive Prostate Cancer
Brief Title: In Men With Metastatic Prostate Cancer, What is the Safety and Benefit of Lutetium-177 PSMA Radionuclide Treatment in Addition to Chemotherapy
Acronym: UpFrontPSMA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Movember Foundation (Other); Prostate Cancer Research Alliance (Unknown); United States Department of Defense (U.S. Federal Agency); Advanced Accelerator Applications (Industry); Australia's Nuclear Science and Technology Organisation (ANSTO) (Unknown); Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Australasian Radiopharmaceutical Trials network (ARTnet) (Unknown); Centre for Biostatistics and Clinical Trials (BaCT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/195
Record Dates: First submitted 2020-04-01; First posted 2020-04-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Hormone Naive Prostate Cancer
MeSH Terms: interventions — Pluvicto; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 177Lu-PSMA+ Docetaxel (Experimental): 7.5 GBq (± 10%) 177Lu-PSMA every 6 weeks x 2 cycles. Docetaxel 75 mg/m2 commencing 6 weeks later, every 3 weeks x 6 cycles
  Interventions: Drug: 177Lu-PSMA-617; Drug: Docetaxel
- Docetaxel (Control) (Other): Docetaxel 75 mg/m2 every 3 weeks x 6 cycles
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Patients will be given 7.5GBq of 177Lu-PSMA every 6 weeks for 2 cycles.
  Other Names: 177Lu-PSMA-617 also referred to as 177Lu-PSMA
  Arms: 177Lu-PSMA+ Docetaxel
Drug: Docetaxel — Docetaxel 75 mg/m2 given every 3 weeks for 6 cycles
  Other Names: Taxotere (trade name)

SUMMARY:
This phase 2 randomised clinical trial will compare the effectiveness of Lu-PSMA therapy followed by docetaxel chemotherapy versus docetaxel chemotherapy on its own in patients with newly-diagnosed high-volume metastatic hormone-naive prostate cancer (mHNPC).

DETAILED DESCRIPTION:
This is an open label, randomised, stratified, 2-Arm, multi-centre, phase 2 clinical trial recruiting 140 newly-diagnosed high-volume mHNPC patients at 11 Australian centres over a period of 18 months. Patients will be randomised to the experimental Arm (177Lu-PSMA followed by docetaxel) or standard-of-care Arm (docetaxel) in a 1:1 ratio. All patients will receive ADT continuously throughout the trial. Patients will be stratified according to disease volume by conventional imaging (low-volume vs. high-volume) and duration of ADT at time of registration (≤ 28 days vs. > 28 days).

ELIGIBILITY:
Inclusion Criteria for study registration:

1. Patient has provided written informed consent
2. Male aged 18 years or older at screening
3. Prostate cancer diagnosed within 12 weeks of commencement of screening
4. Histologically or cytologically confirmed adenocarcinoma of the prostate without significant neuroendocrine differentiation or small cell histology OR metastatic disease typical of prostate cancer (i.e. involving bone or pelvic lymph nodes or para-aortic lymph nodes) with a rising serum PSA
5. Evidence of metastatic disease on CT and/or bone scan
6. PSA > 10ng/ml prior to commencement of medical ADT or surgical orchidectomy
7. Adequate haematological, renal and hepatic functions as defined by:

   * Absolute neutrophil count >1.5 x 109/L
   * Platelet count >100 x 109/L
   * Haemoglobin ≥ 90g/L (no red blood cell transfusion in 4 weeks prior to randomisation)
   * Creatinine Clearance ≥ 40mL/min (Cockcroft-Gault formula)
   * Total bilirubin < 1.5 x ULN (unless known or suspected Gilbert syndrome)
   * Aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 2.0 x ULN (or ≤ 5.0 x ULN in the presence of liver metastases)
8. Have a performance status of 0-2 on the ECOG Performance Scale (see Appendix 1)
9. Life expectancy greater than 6 months with treatment
10. Assessed by a medical oncologist as suitable for treatment with docetaxel
11. Patients must agree to use an adequate method of contraception
12. Willing and able to comply with all study requirements, including all treatments and required assessments including follow-up

Exclusion Criteria for Registration:

1. Any prior pharmacotherapy, radiation therapy, or surgery for metastatic prostate cancer. The following exceptions are permitted:

   * Up to 4 weeks of ADT with luteinising hormone releasing hormone agonists or antagonists or orchiectomy ± concurrent anti-androgens are permitted prior to commencement of screening. At investigator discretion, patients may start ADT at commencement of protocol therapy
   * Up to one course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 14 days prior to registration
2. Symptomatic cord compression, or clinical or imaging findings concerning for impending cord compression
3. Central nervous system metastases
4. Patients with Sjogren's syndrome
5. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
6. Prior diagnosis of another cancer that was:

   * More than 3 years prior to current diagnosis with subsequent evidence of disease recurrence or clinical expectation of recurrence greater than 10%
   * Within 3 years of current diagnosis with the exception of successfully treated basal cell or squamous cell skin carcinoma or adequately treated non-muscle invasive bladder cancer (Tis, Ta and low grade T1 tumours)

Inclusion Criteria for Randomisation:

1. Significant PSMA avidity on 68Ga-PSMA PET/CT, defined after central review as a minimum uptake of SUVmax 15 at a site of disease
2. High-volume metastatic disease on 68Ga-PSMA PET/CT defined as visceral metastases or ≥ 4 bone metastases with ≥ 1 outside the vertebral column and pelvis (extra-axial skeleton)
3. Patient continues to meet all the inclusion criteria for registration

Exclusion Criteria for Randomisation:

1. Major FDG-PET discordance defined as presence of FDG positive disease with minimal PSMA expression in multiple sites (>5) or in more than 50% of total disease volume
2. All the exclusion criteria for registration continue to not apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with a diagnosis of de novo high-volume mHNPC by PSMA-PET/CT criteria
Enrollment: 130 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Undetectable prostate specific antigen (PSA) rate at 12 months after commencement of protocol therapy | Upto 32 months assuming 18 months to complete recruitment, a maximum of 1.6 months from consent to commencement of treatment for last patient and then 12 months from commencement of treatment for last patient.
  Undetectable PSA is defined as PSA ≤ 0.2ng/ml at 12 months after protocol treatment commencement. Patients who experience unequivocal radiographic (by conventional imaging modality) and/or clinical disease progression within 12 months of initiating protocol treatment will be considered as not having undetectable PSA at 12 months.

SECONDARY OUTCOMES:
Safety of 177Lu-PSMA followed by docetaxel compared to docetaxel alone | Through completion of treatment, maximum 26 months.
  The type, grade and relationship to treatment of adverse events (AE) will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0
Time to development of castration resistance between treatment Arms | Through study completion, up until 2 years after the last patient commences treatment.
  Castration resistance is defined as rising PSA and/or radiographic progression despite castrate levels of testosterone (≤ 50ng/dL or ≤ 1.73nmol/L).To be measured from the date of randomisation to the date of first evidence of castration resistance.
PSA-progression free survival (PSA-PFS) between treatment Arms | Through study completion, up until 2 years after the last patient commences treatment.
  PSA progression is defined as a rise in PSA by more than 25% AND more than 2ng/mL above the nadir (lowest PSA point). This needs to be confirmed by a repeat PSA performed at least 3 weeks later. Early rises in PSA prior to 12 weeks will be disregarded in determining PSA progression. To be measured from the date of randomisation to the first date of evidence of PSA progression or date of death due to any cause.
Radiographic-PFS (rPFS) between treatment Arms | Through study completion, up until 2 years after the last patient commences treatment.
  Radiographic progression will be assessed by the investigator per RECIST1.1 for soft tissue and PCWG3 for bone lesions. To be measured from randomisation to the first date of documented radiographic progression using conventional imaging or death due to any cause, whichever occurs first.
Early PSMA PET response between treatment Arms | Through completion of 3 months after treatment commencement for last patient, maximum 23 months.
  PSMA PET response assessed 3 months after treatment commencement defined by central imaging review of 68Ga-PSMA PET CT images.
Describe and compare health-related QoL within 12 months of treatment commencement between treatment Arms | Through completion of 12 months after treatment commencement of last patient, maximum 32 months.
  QoL will be assessed using the Functional Assessment of Cancer Therapy for Prostate Cancer (FACT-P) questionnaire. The primary endpoint for QoL is the area under the curve (AUC) of the trial outcome index (TOI).
  QoL will be assessed at baseline, 6 weeks, 3 months, 6 months, 9 months and 12 months and will be scored according to the respective manuals.
Describe and compare pain within 12 months of treatment commencement between treatment Arms | Through completion of 12 months after treatment commencement of last patient, maximum 32 months.
  Pain will be assessed using the Brief Pain Inventory - Short Form (BPI-SF). The primary endpoint for pain is the area under the curve (AUC) of the worst pain in 24h.
  Pain and QoL will be assessed at baseline, 6 weeks, 3 months, 6 months, 9 months and 12 months and will be scored according to the respective manuals.
Overall survival (OS) between treatment Arms | Through study completion, up until 2 years after the last patient commences treatment.
  OS is defined as the time from randomisation to the date of death due to any cause.

OTHER OUTCOMES:
Assess the correlation between PSMA and FDG PET/CT parameters and clinical outcomes | Through study completion, up until 2 years after the last patient commences treatment.
  Prognostic and predictive value of PET-derived parameters including molecular tumour volume parameters (volume, SUVmax, SUVmean) and radiomics from PET, CT or bone scans using data-characterisation algorithms will be assessed.
Identify biomarkers potentially associated with clinical outcomes | Through study completion, up until 2 years after the last patient commences treatment.
  Prognostic and predictive biomarkers associated with treatment outcome and response will be assessed. This will include any of the following: i) circulating tumour DNA ± tumour tissue (DNA repair genes, tumour suppressor genes, androgen receptor); and ii) whole blood RNA (androgen receptor splice variants, TMPRSS2:ERG fusion).

CONTACTS AND LOCATIONS:
Overall Officials: Arun Azad, MBBS PhD FRACP, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Michael Hofman, MBBS(Hons),FRACP,FAANMS,FICIS, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (12):
- Australia (12):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore, St Leonards, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Cabrini Hospital, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azad AA, Bressel M, Tan H, Voskoboynik M, Suder A, Weickhardt AJ, Guminski A, Francis RJ, Saghebi J, Dhiantravan N, Joshua AM, Emmett L, Horvath L, Murphy DG, Hsiao E, Balakrishnar B, Lin P, Redfern A, Macdonald W, Ng S, Lee ST, Pattison DA, Nadebaum D, Kirkwood ID, Hofman MS; UpFrontPSMA Study Team. Sequential [177Lu]Lu-PSMA-617 and docetaxel versus docetaxel in patients with metastatic hormone-sensitive prostate cancer (UpFrontPSMA): a multicentre, open-label, randomised, phase 2 study. Lancet Oncol. 2024 Oct;25(10):1267-1276. doi: 10.1016/S1470-2045(24)00440-6. Epub 2024 Sep 15. PMID 39293461